CLINICAL TRIAL: NCT06102161
Title: Wedge Resection for Ground-glass Opacity-featured Lung Cancer With Size Less Than 2cm and Consolidation-to-tumor Ratio Between 0.25 to 0.5: a Single-arm, Multi-center, Prospective, Confirmatory Phase III Trial
Brief Title: Wedge Resection for Ground-glass Opacity-featured Lung Cancer (ECTOP-1020)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WGGO
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer; Wedge Resection; Ground-glass Opacity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wedge resection (Experimental): Wedge resection is performed for early-stage lung cancer to remove a wedge-shaped section of lung tissue.
  Interventions: Procedure: Wedge resection

INTERVENTIONS:
Procedure: Wedge resection — Wedge resection is a surgical procedure that is done to remove a wedge-shaped section of lung tissue, usually for treating lung cancer. A wedge resection is less invasive than some of the other surgical options used to remove lung cancer.

SUMMARY:
This is a clinical trial from the Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1020. The goal of this clinical trial is to confirm the therapeutic effect of Wedge resection for ground-glass opacity-featured lung cancer with a size less than 2cm and a consolidation-to-tumor ratio between 0.25 to 0.5.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form and are willing to complete the study according to the plan;
2. Aged from 18 to 80 years old;
3. ECOG equals 0 or 1;
4. Not receiving lung cancer surgery before;
5. Intraoperative or postoperative pathologic diagnosis of lung adenocarcinoma;
6. Single lung nodules with ground-glass dominant or pure ground-glass on CT, or multiple lung nodules with the major lesion being the aforementioned nodules;
7. The nodule has a consolidation-to-tumor ratio (CTR) between 0.25 and 0.5 (including 0.25 and 0.5), and the nodule size is less than or equal to 2 cm;
8. peripheral type of nodes, namely, nodes in the outer 1/3 of the lung field.
9. cT1N0M0 tumors;
10. Complete tumor resection by wedge resection as assessed by the surgeon;
11. Not receiving chemotherapy or radiotherapy before.

Exclusion Criteria:

1. Postoperative pathologic diagnosis of adenocarcinoma in situ or minimally invasive adenocarcinoma.
2. CTR is not between 0.25-0.5 or nodule size greater than 2 cm;
3. Cannot be completely resected by wedge resection;
4. Invasive lung adenocarcinoma or lung malignancy other than lung adenocarcinoma diagnosed cytologically or pathologically;
5. Receiving lung cancer surgery before;
6. Receiving radiotherapy or chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  The event is defined as the death due to any causes.

SECONDARY OUTCOMES:
5-year recurrence-free survival | 5 years
  The event is defined as the tumor recurrence.
Postoperative lung function (FEV1) | 5 years
  forced expiratory volume in one second (FEV1)
Postoperative lung function | 5 years
  forced vital capacity (FVC)
Sites of tumor recurrence and metastasis | 5 years
Radical wedge resection (R0 resection) completion rate | 5 years
Surgery-related complications | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li T, Fu F, Zhang Y, Chen H. Protocol for a single-arm, multicenter, prospective, confirmatory phase III trial of wedge resection for invasive ground glass opacity-featured lung cancer with a size </=2 cm and a consolidation tumor ratio between 0.25 and 0.5 (ECTOP-1020 study). J Thorac Dis. 2024 Jul 30;16(7):4711-4718. doi: 10.21037/jtd-24-440. Epub 2024 Jul 9. PMID 39144343